CLINICAL TRIAL: NCT01380743
Title: An Open-Label, Multi-Center, International Study to Investigate Drug-Drug Interactions Between AT2220 and Alglucosidase Alfa in Patients With Pompe Disease
Brief Title: Drug-drug Interaction Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT2220-010
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Pompe Disease
Keywords: Amicus Therapeutics; duvoglustat; AT2220; alpha-glucosidase; alglucosidase alfa
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — 1-Deoxynojirimycin; GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1, Duvoglustat 50 mg + rhGAA (Experimental): During Period 1, participants received a single intravenous infusion of rhGAA. During Period 2, each participant received a single 50 milligram (mg) oral dose of duvoglustat 1 hour prior to initiation of a single rhGAA infusion.
  Participants were on a stable regimen and dose of rhGAA for at least 3 months before screening.
  Interventions: Drug: duvoglustat; Drug: rhGAA
- Cohort 2, Duvoglustat 100 mg + rhGAA (Experimental): During Period 1, participants received a single intravenous infusion of rhGAA. During Period 2, each participant received a single 100 mg oral dose of duvoglustat 1 hour prior to initiation of a single rhGAA infusion.
  Participants were on a stable regimen and dose of rhGAA for at least 3 months before screening.
  Interventions: Drug: duvoglustat; Drug: rhGAA
- Cohort 3, Duvoglustat 250 mg + rhGAA (Experimental): During Period 1, participants received a single intravenous infusion of rhGAA. During Period 2, each participant received a single 250 mg oral dose of duvoglustat 1 hour prior to initiation of a single rhGAA infusion.
  Participants were on a stable regimen and dose of rhGAA for at least 3 months before screening.
  Interventions: Drug: duvoglustat; Drug: rhGAA
- Cohort 4, Duvoglustat 600 mg + rhGAA (Experimental): During Period 1, participants received a single intravenous infusion of rhGAA. During Period 2, each participant received a single 600 mg oral dose of duvoglustat 1 hour prior to initiation of a single rhGAA infusion.
  Participants were on a stable regimen and dose of rhGAA for at least 3 months before screening.
  Interventions: Drug: duvoglustat; Drug: rhGAA

INTERVENTIONS:
Drug: duvoglustat — Single oral dose
  Other Names: AT2220; duvoglustat hydrochloride
Drug: rhGAA — Single intravenous infusion
  Other Names: alglucosidase alfa; recombinant human alpha-glucosidase; Myozyme; Lumizyme

SUMMARY:
This study evaluates drug-drug interactions between AT2220 (duvoglustat) and recombinant human alpha-glucosidase (rhGAA, also known as alglucosidase alfa) in participants with Pompe Disease.

DETAILED DESCRIPTION:
This was a multi-center, international, open-label, two-period, fixed-sequence crossover study to evaluate the safety and pharmacokinetic effect of single ascending doses of duvoglustat on rhGAA administered 1 hour before initiation of a single rhGAA infusion. During Period 1, participants received a single intravenous infusion of rhGAA. During Period 2, each participant received a single oral dose of duvoglustat 1 hour prior to initiation of a single rhGAA infusion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, diagnosed with Pompe disease and between 18 and 65 years of age, inclusive
* Participant has been on a stable regimen and dose of rhGAA for at least 3 months before screening (stable regimen defined as currently receiving rhGAA every 2 weeks and stable dose defined as not varying by more than ± 10%)
* Participant has an estimated glomerular filtration rate (eGFR) ≥ 50 mL/min at Screening; eGFR to be estimated using the 4-parameter Modification of Diet in Renal Disease (MDRD) equation:

eGFR (mL/min/1.73 m^2) = 175 x (Scr)^(-1.154) x (Age)^(-0.203) x (0.742 if female) x (1.212 if African-American)

* Male and female participants of childbearing potential agree to use medically accepted methods of contraception during the study and for 30 days after study completion
* Participant is willing and able to provide written informed consent and is able to comply with all study procedures

Exclusion Criteria:

* Participant has had a documented transient ischemic attack, ischemic stroke, unstable angina, or myocardial infarction within the 3 months before Screening
* Participant has clinically significant unstable cardiac disease (for example, cardiac disease requiring active management, such as symptomatic arrhythmia, unstable angina, or New York Heart Association class III or IV congestive heart failure)
* Participant requiring mechanical ventilation or is confined to a wheelchair
* Participant has a history of allergy or sensitivity to study drug (including excipients) or other iminosugars (for example, miglustat, miglitol)
* Participant is pregnant or breastfeeding
* Participant tests positive for hepatitis B surface antigen or hepatitis C antibody
* Participant has received any investigational/experimental drug or device within 30 days of Screening
* Participant has any intercurrent illness or condition that may preclude the participant from fulfilling the protocol requirements or suggests to the investigator that the potential participant may have an unacceptable risk by participating in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2013-01-04 (Actual); Study Completion 2013-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Study Sponsor (Amicus Therapeutics, Inc)
Locations (15):
- United States (11):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Orange, California
  - Gainesville, Florida
  - Decatur, Georgia
  - Kansas City, Kansas
  - Great Falls, Montana
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
  - Springfield, Virginia
- Hamilton, Ontario, Canada
- Paris, France
- United Kingdom (2):
  - London, Queen Square
  - Salford

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 27 participants were enrolled; 25 participants completed the study. Two participants were discontinued from the study prior to assignment to a cohort: 1 participant voluntarily withdrew before receiving study drug; 1 participant was screened twice and enrolled once, and was counted twice under the total number enrolled.
Groups:
- Cohort 1, Duvoglustat 50 mg + rhGAA: During Period 1, participants received a single intravenous infusion of rhGAA. During Period 2, each participant received a single 50 mg oral dose of duvoglustat 1 hour prior to initiation of a single rhGAA infusion.
- Cohort 2, Duvoglustat 100 mg + rhGAA: During Period 1, participants received a single intravenous infusion of rhGAA. During Period 2, each participant received a single 100 mg oral dose of duvoglustat 1 hour prior to initiation of a single rhGAA infusion.
- Cohort 3, Duvoglustat 250 mg + rhGAA: During Period 1, participants received a single intravenous infusion of rhGAA. During Period 2, each participant received a single 250 mg oral dose of duvoglustat 1 hour prior to initiation of a single rhGAA infusion.
- Cohort 4, Duvoglustat 600 mg + rhGAA: During Period 1, participants received a single intravenous infusion of rhGAA. During Period 2, each participant received a single 600 mg oral dose of duvoglustat 1 hour prior to initiation of a single rhGAA infusion.
Period: Overall Study
Arm/Group | Cohort 1, Duvoglustat 50 mg + rhGAA | Cohort 2, Duvoglustat 100 mg + rhGAA | Cohort 3, Duvoglustat 250 mg + rhGAA | Cohort 4, Duvoglustat 600 mg + rhGAA
Started | 6 | 6 | 6 | 7
Received at Least 1 Dose of Study Drug | 6 | 6 | 6 | 7
Completed | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled and received at least 1 dose of rhGAA or duvoglustat.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Duvoglustat 50 mg + rhGAA | Cohort 2, Duvoglustat 100 mg + rhGAA | Cohort 3, Duvoglustat 250 mg + rhGAA | Cohort 4, Duvoglustat 600 mg + rhGAA | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (5.35) | 52.8 (5.71) | 50.0 (12.90) | 40.0 (6.61) | 47.3 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 2 | 12
  Male | 3 | 3 | 2 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Severe Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event (AE) with an onset date on or after the first dose of investigational medicinal product (IMP), or an AE with an onset date before the first dose date that worsened in severity after the first dose date. A severe AE was defined as an AE that was incapacitating and required medical intervention. The number of participants who experienced 1 or more severe TEAEs after dosing on Day 1 up to Day 60 (includes end of study follow-up period) is reported.
  A summary of serious and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Day 1 after dosing up to Day 60
Population: The Safety Population included all participants who were enrolled and received at least 1 dose of rhGAA or duvoglustat.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Duvoglustat 50 mg + rhGAA | Cohort 2, Duvoglustat 100 mg + rhGAA | Cohort 3, Duvoglustat 250 mg + rhGAA | Cohort 4, Duvoglustat 600 mg + rhGAA
Number analyzed (Participants) | 6 | 6 | 6 | 7
Participants | 0 | 0 | 0 | 1

2. Primary Outcome: Pharmacokinetics (PK): Maximum Measured Plasma Concentration (Cmax) Of Total GAA And rhGAA Protein In Plasma In Participants With Pompe Disease
Description: The Cmax of total GAA and rhGAA protein in plasma was measured after a single rhGAA intravenous infusion and after pre-administration of single ascending oral doses of duvoglustat.
  During Treatment Period 1, participants received a single intravenous infusion of rhGAA. During Treatment Period 2, participants received a single oral dose of duvoglustat 1 hour before initiation of a single rhGAA intravenous infusion. PK samples were taken at time points Predose, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, and 24 hours, and 3 or 7 days postdose during Periods 1 and 2, and 24 to 30 days postdose during Period 2.
Time Frame: Predose, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, and 24 hours, and 3 or 7 days postdose during Periods 1 and 2, and 24 to 30 days postdose during Period 2
Population: The Per Protocol population included all participants who successfully completed both periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/mL/h
Arm/Group | Cohort 1, Duvoglustat 50 mg + rhGAA | Cohort 2, Duvoglustat 100 mg + rhGAA | Cohort 3, Duvoglustat 250 mg + rhGAA | Cohort 4, Duvoglustat 600 mg + rhGAA
Number analyzed (Participants) | 6 | 6 | 6 | 7
nmol/mL/h
  Total GAA, Period 1 | 17269 (25.6) | 22785 (18.1) | 18986 (19.5) | 18980 (34.6)
  Total GAA, Period 2 | 20539 (21.2) | 28607 (14.1) | 22651 (9.0) | 22989 (36.4)
  rhGAA, Period 1 | 328660 (40.7) | 399622 (33.2) | 405543 (11.4) | 507294 (47.9)
  rhGAA, Period 2 | 385475 (35.7) | 430738 (39.5) | 438795 (7.0) | 637571 (48.8)

3. Primary Outcome: PK: Time To The Maximum Plasma Concentration (Tmax) Of Total GAA And rhGAA Protein In Plasma In Participants With Pompe Disease
Description: The Tmax of total GAA and rhGAA protein in plasma was measured after a single rhGAA intravenous infusion and after pre-administration of single ascending oral doses of duvoglustat.
  During Treatment Period 1, participants received a single intravenous infusion of rhGAA. During Treatment Period 2, participants received a single oral dose of duvoglustat 1 hour before initiation of a single rhGAA intravenous infusion. PK samples were taken at time points Predose, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, and 24 hours, and 3 or 7 days postdose during Periods 1 and 2, and 24 to 30 days postdose during Period 2.
Time Frame: as for outcome 2
Population: The Per Protocol population included all participants who successfully completed both periods.
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1, Duvoglustat 50 mg + rhGAA | Cohort 2, Duvoglustat 100 mg + rhGAA | Cohort 3, Duvoglustat 250 mg + rhGAA | Cohort 4, Duvoglustat 600 mg + rhGAA
Number analyzed (Participants) | 6 | 6 | 6 | 7
h
  Total GAA, Period 1 | 4.74 [4.00 to 5.00] | 4.00 [2.98 to 4.97] | 4.00 [3.78 to 4.02] | 4.00 [3.00 to 6.00]
  Total GAA, Period 2 | 4.51 [3.95 to 5.98] | 4.00 [3.00 to 5.98] | 4.00 [4.00 to 4.00] | 4.00 [3.00 to 6.00]
  rhGAA, Period 1 | 4.98 [4.00 to 5.00] | 4.01 [4.00 to 5.07] | 4.01 [3.78 to 5.00] | 4.00 [3.83 to 6.00]
  rhGAA, Period 2 | 4.98 [4.00 to 6.02] | 4.00 [4.00 to 7.00] | 4.50 [4.00 to 7.02] | 4.00 [3.00 to 6.00]

4. Primary Outcome: PK: Elimination Half-life (T1/2) Of Total GAA And rhGAA Protein In Plasma In Participants With Pompe Disease
Description: The T1/2 of total GAA and rhGAA protein in plasma was measured after a single rhGAA intravenous infusion and after pre-administration of single ascending oral doses of duvoglustat.
  During Treatment Period 1, participants received a single intravenous infusion of rhGAA. During Treatment Period 2, participants received a single oral dose of duvoglustat 1 hour before initiation of a single rhGAA intravenous infusion. PK samples were taken at time points Predose, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, and 24 hours, and 3 or 7 days postdose during Periods 1 and 2, and 24 to 30 days postdose during Period 2.
  Values presented are arithmetic mean (percent coefficient of variation, [CV%]). The number of participants analyzed for some cohorts are reduced because the terminal phase of the concentration profile for these participants was not estimable.
Time Frame: as for outcome 2
Population: The Per Protocol population included all participants who successfully completed both periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Cohort 1, Duvoglustat 50 mg + rhGAA | Cohort 2, Duvoglustat 100 mg + rhGAA | Cohort 3, Duvoglustat 250 mg + rhGAA | Cohort 4, Duvoglustat 600 mg + rhGAA
Number analyzed (Participants) | 6 | 6 | 6 | 7
h
  Total GAA, Period 1 | 3.81 (12.7) | 3.82 (17.7) | 3.56 (13.7) | 3.70 (19.9)
  Total GAA, Period 2 | 4.42 (16.9) | 4.77 (14.2) | 5.36 (26.0) | 6.33 (22.8)
  rhGAA, Period 1: number analyzed (Participants) | 6 | 5 | 6 | 4
  rhGAA, Period 1 | 3.31 (39.6) | 2.33 (59.5) | 1.89 (46.9) | 2.33 (54.3)
  rhGAA, Period 2: number analyzed (Participants) | 6 | 4 | 6 | 7
  rhGAA, Period 2 | 4.43 (38.1) | 5.76 (55.6) | 4.23 (52.3) | 5.71 (45.6)

5. Primary Outcome: PK: Area Under The Plasma Concentration Versus Time Curve From Time 0 To The Time Of The Last Measurable Concentration (AUC0-t) Of Total GAA And rhGAA Protein In Plasma In Participants With Pompe Disease
Description: The AUC0-t of total GAA and rhGAA protein in plasma was measured after a single rhGAA intravenous infusion and after pre-administration of single ascending oral doses of duvoglustat.
  During Treatment Period 1, participants received a single intravenous infusion of rhGAA. During Treatment Period 2, participants received a single oral dose of duvoglustat 1 hour before initiation of a single rhGAA intravenous infusion. PK samples were taken at time points Predose, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, and 24 hours, and 3 or 7 days postdose during Periods 1 and 2, and 24 to 30 days postdose during Period 2.
Time Frame: as for outcome 2
Population: The Per Protocol population included all participants who successfully completed both periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/mL/h
Arm/Group | Cohort 1, Duvoglustat 50 mg + rhGAA | Cohort 2, Duvoglustat 100 mg + rhGAA | Cohort 3, Duvoglustat 250 mg + rhGAA | Cohort 4, Duvoglustat 600 mg + rhGAA
Number analyzed (Participants) | 6 | 6 | 6 | 7
nmol/mL/h
  Total GAA, Period 1 | 108578 (24.1) | 141515 (27.9) | 107489 (21.7) | 118483 (43.1)
  Total GAA, Period 2 | 159994 (18.1) | 226198 (25.4) | 201044 (8.3) | 228413 (38.4)
  rhGAA, Period 1 | 1891079 (35.6) | 2227356 (62.8) | 2248866 (24.7) | 2326168 (55.5)
  rhGAA, Period 2 | 2914884 (49.2) | 3466263 (59.5) | 3618948 (26.4) | 5293233 (68.2)

6. Primary Outcome: PK: AUC From Time 0 Extrapolated To Infinity (AUCinf) Of Total GAA And rhGAA Protein In Plasma In Participants With Pompe Disease
Description: The AUCinf of total GAA and rhGAA protein in plasma was measured after a single rhGAA intravenous infusion and after pre-administration of single ascending oral doses of duvoglustat.
  During Treatment Period 1, participants received a single intravenous infusion of rhGAA. During Treatment Period 2, participants received a single oral dose of duvoglustat 1 hour before initiation of a single rhGAA intravenous infusion. PK samples were taken at time points Predose, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, and 24 hours, and 3 or 7 days postdose during Periods 1 and 2, and 24 to 30 days postdose during Period 2.
  The number of participants analyzed for some cohorts are reduced because the terminal phase of the concentration profile for these participants was not estimable.
Time Frame: as for outcome 2
Population: The Per Protocol population included all participants who successfully completed both periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*(nmol/mL/h)
Arm/Group | Cohort 1, Duvoglustat 50 mg + rhGAA | Cohort 2, Duvoglustat 100 mg + rhGAA | Cohort 3, Duvoglustat 250 mg + rhGAA | Cohort 4, Duvoglustat 600 mg + rhGAA
Number analyzed (Participants) | 6 | 6 | 6 | 7
h*(nmol/mL/h)
  Total GAA, Period 1 | 110388 (24.5) | 144056 (28.6) | 108862 (22.1) | 120604 (44.3)
  Total GAA, Period 2 | 165983 (19.1) | 237613 (27.6) | 215276 (9.5) | 254074 (42.0)
  rhGAA, Period 1: number analyzed (Participants) | 6 | 5 | 6 | 4
  rhGAA, Period 1 | 2274897 (35.5) | 2232099 (54.0) | 2468980 (26.4) | 2452414 (70.5)
  rhGAA, Period 2: number analyzed (Participants) | 6 | 3 | 6 | 7
  rhGAA, Period 2 | 3603068 (37.4) | 3427088 (71.1) | 4602726 (31.3) | 6691323 (46.6)

7. Secondary Outcome: Total GAA Activity In Skeletal Muscle
Description: The total GAA activity in skeletal muscle was measured after a single intravenous administration of rhGAA alone and after pre-administration of single ascending oral doses of duvoglustat. Participants were assessed using skeletal muscle biopsies at either Day 3 or Day 7 during Treatment Periods 1 and 2.
Time Frame: Day 3 or Day 7
Population: The Per Protocol population included all participants who successfully completed both periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/mg/h
Arm/Group | Cohort 1, Duvoglustat 50 mg + rhGAA | Cohort 2, Duvoglustat 100 mg + rhGAA | Cohort 3, Duvoglustat 250 mg + rhGAA | Cohort 4, Duvoglustat 600 mg + rhGAA
Number analyzed (Participants) | 6 | 6 | 6 | 6
pmol/mg/h
  Total GAA, Period 1, Day 3: number analyzed (Participants) | 2 | 3 | 3 | 3
  Total GAA, Period 1, Day 3 | 1409 (130) | 1926 (67) | 2622 (14) | 1887 (47)
  Total GAA, Period 2, Day 3: number analyzed (Participants) | 2 | 3 | 3 | 3
  Total GAA, Period 2, Day 3 | 1952 (8) | 2320 (77) | 2746 (35) | 2710 (37)
  Total GAA, Period 1, Day 7: number analyzed (Participants) | 4 | 3 | 3 | 3
  Total GAA, Period 1, Day 7 | 1216 (24) | 861 (16) | NA (91) — Value not calculated because 1 participant's value was below the limit of quantification. | 916 (25)
  Total GAA, Period 2, Day 7: number analyzed (Participants) | 4 | 3 | 3 | 3
  Total GAA, Period 2, Day 7 | 1197 (18) | 1064 (39) | 1690 (22) | 1085 (14)

8. Secondary Outcome: Duvoglustat Concentration In Skeletal Muscle
Description: The concentration of duvoglustat in skeletal muscle tissue homogenate was measured after pre-administration of single ascending oral doses of duvoglustat during Treatment Period 2. Participants had skeletal muscle biopsies at either Day 3 or Day 7 during Treatment Period 2.
  Three participants were excluded from this analysis due to the following reasons: treatment sequence was inadvertently switched due to study site error, follow-up biopsy sample could not be conclusively identified, or muscle biopsies were mislabeled at the clinical site.
  Values presented are arithmetic mean (percent coefficient of variation, [CV%]) because of the prevalence of participants with values below the limit of quantification. Concentrations below the limit of quantification were treated as zero.
Time Frame: Day 3 or Day 7
Population: The Per Protocol population included all participants who successfully completed both periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/g
Arm/Group | Cohort 1, Duvoglustat 50 mg + rhGAA | Cohort 2, Duvoglustat 100 mg + rhGAA | Cohort 3, Duvoglustat 250 mg + rhGAA | Cohort 4, Duvoglustat 600 mg + rhGAA
Number analyzed (Participants) | 6 | 6 | 6 | 7
ng/g
  Duvoglustat Concentration, Day 3: number analyzed (Participants) | 1 | 3 | 3 | 1
  Duvoglustat Concentration, Day 3 | 0 (NA) — Value was not calculated because participant's value was below the limit of quantification. | 5.9 (173) | 38.8 (87) | 83.6 (NA) — Value was not calculated because participant's value was below the limit of quantification.
  Duvoglustat Concentration, Day 7: number analyzed (Participants) | 4 | 3 | 2 | 3
  Duvoglustat Concentration, Day 7 | 8.7 (68) | 0 (NA) — Value was not calculated because participant's value was below the limit of quantification. | 28.0 (0.5) | 54.1 (25)

ADVERSE EVENTS:
Time Frame: Day 1 after dosing up to Day 60
Arm/Group | Cohort 1, Duvoglustat 50 mg + rhGAA | Cohort 2, Duvoglustat 100 mg + rhGAA | Cohort 3, Duvoglustat 250 mg + rhGAA | Cohort 4, Duvoglustat 600 mg + rhGAA
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 5/6 | 3/6 | 4/6 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Duvoglustat 50 mg + rhGAA (N=6) | Cohort 2, Duvoglustat 100 mg + rhGAA (N=6) | Cohort 3, Duvoglustat 250 mg + rhGAA (N=6) | Cohort 4, Duvoglustat 600 mg + rhGAA (N=7)
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cohort 1, Duvoglustat 50 mg + rhGAA (N=6) | Cohort 2, Duvoglustat 100 mg + rhGAA (N=6) | Cohort 3, Duvoglustat 250 mg + rhGAA (N=6) | Cohort 4, Duvoglustat 600 mg + rhGAA (N=7)
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Uterine enlargement (Reproductive system and breast disorders) | 0/3 | 0/3 | 0/4 | 1/2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can only publish the results from this trial provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review. If requested, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.